CLINICAL TRIAL: NCT02261610
Title: Interest of PCT in the Management of Antibiotic for the Patient With a Febrile Pulmonary Embolism.
Brief Title: Pulmonary Embolism and PCT. PE-PCT Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty of recrutement
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0203; 2014-A00046-41
Record Dates: First submitted 2014-09-05; First posted 2014-10-10 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Embolism With Fever
Keywords: PCT algorithm; Antibiotic; Pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism

ARMS (2):
- clinical group (Experimental): In the first group of patients, the use of antibiotics will be guided by clinical (clinical group).
  Interventions: Procedure: Procalcitonin algorithm
- PCT group (Other): In the second group, the use of antibiotics will be guided by the algorithm (PCT group).
  Interventions: Procedure: Procalcitonin algorithm

INTERVENTIONS:
Procedure: Procalcitonin algorithm — Procalcitonin algorithm (usually used for lower respiratory tract) guide antibiotic therapy

SUMMARY:
The clinical manifestations of pulmonary embolism vary greatly from the absence of specific clinical symptoms to cardiogenic shock or cardiac arrest. Clinical form of EP represented by "lung superinfection", also called "pulmonary embolism superinfected" is common and represents up to 30% of initial clinical presentations; she been few evaluations in clinical research. The reality of the bacterial infection remains controversial and the clinical presentation often leads to the prescription of empirical antibiotic therapy, often unnecessary in many cases. Number of antibiotic prescriptions are probably inappropriate.

Fever has long been recognized as a sign associated with pulmonary embolism. Stein et al reported a temperature above 37.5 ° C on 50% of patients with acute pulmonary embolism without actually clarified whether this was related to temperature with a pulmonary embolism or other associated cause. Murray et al estimated that greater than 38 ° C was explained by pulmonary embolism in 57.1% of patients while in the PIOPED study, only 14% of patients had fever with no other cause identified as pulmonary embolism. Fever due to pulmonary embolism is often low intensity (often less than 38.3) and of short duration, with a peak on the day of pulmonary embolism and a gradual decrease of about 1 week. The pathophysiology of fever in pulmonary embolism has not yet was completely clarified. It is suggested that a combination of several factors involved pyrogenic myocardial tissue necrosis and releasing pro-inflammatory cytokines, hemorrhage, vascular irritation or inflammation, atelectasis or local superinfection.

Since 2004, the PCT has become a marker helping the initiation of antibiotic therapy in patients with community-acquired pneumonia. This is especially verified in patients admitted for acute exacerbation of chronic obstructive bronchitis. In the latter case, the use of PCT reduces inappropriate antibiotic prescribing. Thus helping the clinician by measuring biomarkers such as PCT is based on writing an algorithm leading or not to use antibiotics.

The use of an algorithm involving the PCT could just as for infectious pneumonia or COPD, of interest in the febrile pulmonary embolism to distinguish febrile forms related to bacterial infections febrile forms of EP to other causes.

DETAILED DESCRIPTION:
The investigators propose to realize a single-center prospective, randomized, parallel group, to compare two groups of patients admitted with febrile pulmonary embolism . In the first group of patients, the use of antibiotics will be guided by clinical (clinical group). In the second group, the use of antibiotics will be guided by the algorithm (PCT group). The guided by the PCT algorithm is only given aid the clinician in the therapeutic management without its application only requires the doctor in charge of the patient. So if your doctor may advocate (or deemed necessary) to continue (or start) antibiotics even if the PCT algorithm would allow him to stop (or not initiate).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* CT diagnosis of pulmonary embolism
* Temperature> 37.8 ° C
* About affiliated to the social security
* Prior agreement with the patient signing a consent

Exclusion Criteria:

* Pregnant Woman
* Refusal of the patient
* Pulmonary Neoplasia
* Antibiotic ongoing for more than 24 hours at the time of diagnosis of pulmonary embolism
* Cardiogenic shock (hypotension with mean arterial pressure less than 65 bpm)
* Suspicion of infection other than lung associated (associated urinary tract infection, prostatitis, ENT infection, sinusitis ...)
* Patient under guardianship
* Patients unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-11-24 (Actual)

PRIMARY OUTCOMES:
Percentage of patient treated by antibiotics in each group | at day 1

SECONDARY OUTCOMES:
Percentage of death | at day 1
Percentage of antibiotics stop | at day 1
Rate of new hospitalization during the following month | at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Farès MOUSTAFA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France